CLINICAL TRIAL: NCT03300375
Title: Exercise Intervention for Unilateral Amputees With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201701256; OCR18330 (Other: University of Florida)
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Two group, parallel study
Who Masked: Participant
Masking Description: Permuted block randomization with block sizes of four will made by means of a computer algorithm to ensure balanced group sizes and allocation concealment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-Based Resistance Exercise Intervention Group (Active Comparator): Participants in the HBRX group will be coached through six phases of the intervention with two weeks per phase. Exercise will use body weight and resistance exercise bands. A set of commercial elastic resistive bands and a stability pad (TheraBand, Inc.) will be provided to each participant to keep for personal use after their participation in the study. The use of elastic bands for resistance training can induce similar results in neuromuscular adaptations as well as strength to those achieved by weight machines and free-weights.
  Interventions: Other: Home exercise program
- Wait-List Control Condition Group (Experimental): Participants who are assigned to the CON group will wait to participate in the resistance training after a three month wait period. Participants will follow all instructions provided to them by their physician and care team, but will be asked to refrain from starting any new strengthening exercise protocols or begin any new physical therapies during this time. The participants will be contacted by phone on a monthly basis during the study period to determine if any changes in LBP symptoms have occurred. At month three, these participants will also receive the elastic resistive bands and a stability pad.
  Interventions: Other: Home exercise program; Other: Post Op instructions

INTERVENTIONS:
Other: Home exercise program — Home-based, progressive exercise program using resistance bands
Other: Post Op instructions — Participants will follow all instructions provided to them by their physician and care team, but will be asked to refrain from starting any new strengthening exercise protocols or begin any new physical therapies during this time.
  Arms: Wait-List Control Condition Group

SUMMARY:
A three-month, randomized, controlled study will be used to examine the effects of a home-based resistance exercise program on improving pain severity and functional ability in unilateral lower extremity amputees who suffer from Low Back Pain. The study will follow the principles of the Consolidated Standards of Reporting Trials for randomized, two group, parallel studies.

DETAILED DESCRIPTION:
Amputation to the lower extremity is a life-changing event. Approximately 2 million Americans live with limb loss, with ~45% of losses occurring from traumatic mechanisms. After the injury has healed and a prosthetic limb is fitted, the long-term care for amputees typically focuses on maintenance of the prosthesis fit and optimizing physical function. Even with high-quality prostheses, amputation permanently impacts biomechanical symmetry of gait. After unilateral transtibial or transfemoral amputation, skeletal muscle atrophy occurs in the lower extremity and back. Asymmetric gait causes mechanical stresses at lumbar spine, and loss of muscle mass and strength, all of which exaggerate gait aberrations. As a result, chronic low back pain (LBP) can develop. LBP is a common, but often unaddressed, secondary complication in over half of the unilateral amputee population.

Lower extremity amputees face numerous physical and emotional challenges after their injuries. Performing ambulatory activities are more physically demanding with an amputation than without. The psychological stress levels are often high after an amputation, contributing to activity avoidance and limiting participation in load-bearing activities. LBP independently contributes to costly health burdens such as addiction to pain medicine, depression and lifestyle diseases and LBP erodes physical and mental quality of life (QOL). Pain is also related to skeletal muscle atrophy in the low back. The combination of an amputation injury and LBP may amplify ambulation-related limitations and further deteriorate QOL. Unilateral lower extremity amputees who suffer from chronic LBP therefore may therefore experience greater walking limitations, physical activity avoidance and physiological changes to skeletal muscle, strength and perceived QOL than people with back pain or amputation alone.

Long-term care for amputees requires a team of physicians, prostheticians, therapists and other specialists. Patients often travel long distances to receive their care. Patients with limited resources may not be able to maintain a long-term relationship with therapists due to cost restrictions. Home-based interventions that target LBP could substantially impact the secondary disease burden and help restore QOL in the amputee population. In the general population, evidence indicates that consistently-performed muscle strengthening activity is associated with significantly lower odds of developing back pain in men and women. Resistance exercise is effective for lumbar muscle strength gains, functional gains in ambulation and movement and for improving both physical and mental aspects of QOL. Resistance training benefits in strength, motor skills, and many aspects of quality of life (both functional and psychosocial) are seen throughout several different demographics; from young adults to the elderly.

Current clinical paradigms to treat general LBP include referral to physical therapy for strengthening exercise programs. For amputees, challenges to receiving therapeutic care include travel distance, and financial limitations for exercise facility memberships or therapy copayments. Patients may not be able to sustain and therapy gains over the long-term when therapy benefits run out. Thus, exercise to treat LBP in amputees must be accessible, low or no cost and sustainable. A significant deficit in the clinical literature is that the study team does not know the effectiveness of home-based resistance training on different chronic musculoskeletal pains in amputees. Moreover, the mechanisms that may contribute to effectiveness of strength training on pain relief in amputees are not clear. The problem is therefore multifaceted: 1) amputees experience permanent anatomic changes that impact load-bearing activity, back pain and QOL; 2) chronic LBP treatment is not often a focus for the long-term management of the unilateral lower extremity amputee; 3) chronic LBP can develop in amputees as a consequence of asymmetric movement patterns, lumbar muscle atrophy and low muscle strength, but the relative contribution of each to pain severity is not known. These evidence gaps are significant barriers to the optimization of care for this special population by clinical teams who care for these individuals, and for determination of pain responders with strengthening exercise.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-60 years of age
* English speaking
* Suffering from chronic LBP (>3 months with ≥3 pain episodes per week)
* Baseline pain of ≥3 points out of 10 on the NRSPain scale
* Amputation ≥1 year prior and their current prosthesis must have been worn for at least 6 months (prosthesis K-Level of K2 or greater, indicating the subject is able to ambulate and traverse low-level environmental barriers such as curbs, stairs, or uneven surfaces).
* Must have regular access to a computer for skype, or a mobile phone or iPAD to perform facetime

Exclusion Criteria:

* Acute back injury
* Any other chronic back pathology (i.e. herniated disc, ankylosing spondylosis, other related neurologic disease)
* Pain symptoms or functional limitations (including those that may require assistive devices) that preclude participation in resistance exercise or physical activity
* Back surgery within the past two years that restrict daily physical activities
* Currently enrolled in any other resistance or strengthening exercise interventions
* Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Up to 6 months
  Pain and Catastrophizing Scale (PCS) is a 13 item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). The PCS is broken into three subscales being magnification, rumination, and helplessness. The scale was developed as a self-report measurement tool that provided a valid index of catastrophizing in clinical and non-clinical populations.
Functional impairment due to back pain | Up to 6 months
  Roland Disability Questionnaire consist of 24 items (see below). Those 24 questions are related specifically to physical functions that were likely to be affected by low back pain. Greater levels of disability are reflected by higher numbers. Scores under 4 and over 20 may not show significant change over time in patients with scores of less than 4 and deterioration in patients who have scores greater than 20.
Quality of Life Assessment | Up to 6 months
  Medical Outcomes Short-Form 36 (SF-36) This instrument has 36 items and yields eight domain scores and two component scores (Mental, Physical). The eight domains are: physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems and emotional well-being. The SF-36 has shown good internal consistency (Cronbach's range of 0.95-0.93). This instrument has been used to track QOL after traumatic injury, such as amputation.50

SECONDARY OUTCOMES:
Functional disability in patients with low back pain | up to 6 months
  Oswestry Disability Questionnaire: 0-20% Minimal disability; 20-40% Moderate disability; 40-60% Severe disability; 60-80% Crippled; 80-100% bed-bound.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Vincent, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wasser JG, Herman DC, Horodyski M, Zaremski JL, Tripp B, Page P, Vincent KR, Vincent HK. Exercise intervention for unilateral amputees with low back pain: study protocol for a randomised, controlled trial. Trials. 2017 Dec 29;18(1):630. doi: 10.1186/s13063-017-2362-0. PMID 29284521